CLINICAL TRIAL: NCT06161454
Title: A Feasibility Study of Xofluza Treatment of Influenza in Pediatric Transplant Recipients, Waitlisted Subjects and Household Members After Early Infection Alerting Using Wearable Devices
Brief Title: Xofluza-Wearables Feasibility-Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-020440
Record Dates: First submitted 2023-11-27; First posted 2023-12-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Infection, Coronavirus; Infections; Influenza; Transplant; Infection Viral
Keywords: Transplant; Infections; Wearable Devices; smart wearable device; Xofluza; Influenza
MeSH Terms: conditions — Coronavirus Infections; Infections; Influenza, Human; Virus Diseases | interventions — baloxavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Population 1: Transplant Recipients (Experimental): Participants who are a CHOP kidney, heart, liver or lung single or multiple transplant recipients aged 5 years or older will receive a single dose of Baloxavir.
  Interventions: Drug: Baloxavir Marboxil
- Population 2: Waitlisted Patients for Transplant (Experimental): Participants who are waitlisted CHOP kidney, heart, liver or lung single or multiple transplant recipients aged 5 years or older will receive a single dose of Baloxavir marboxil.
  Interventions: Drug: Baloxavir Marboxil
- Population 3: Household Members (Non-Transplant) (Experimental): Non-Transplanted Household Members aged 5 years or older will receive a single dose of Baloxavir marboxil.
  Interventions: Drug: Baloxavir Marboxil
- Population 4: Non-Baloxavir treatment subjects (No Intervention): CHOP transplant recipients and all other non-transplanted household members who are 2-4 years of age.
  Subjects 5 years and up who are Influenza positive but whom do not receive Baloxavir treatment

INTERVENTIONS:
Drug: Baloxavir Marboxil — Baloxavir marboxil will be administered as either a tablet or granules. Dose is based on body weight:
  40 mg for a participants weighing 20-79 kg, or 80 mg for a patient weighing more than or equal to 80 kg
  Other Names: Xofluza
  Arms: Population 1: Transplant Recipients; Population 2: Waitlisted Patients for Transplant; Population 3: Household Members (Non-Transplant)

SUMMARY:
The goal of this prospective, interventional, single-center study is to assess whether the early detection of Influenza with smart wearable device algorithms and alerting, rapid testing, and subsequent Baloxavir treatment demonstrate better post-infection outcomes versus publicly available- and Centers for Disease Control (CDC)-derived national statistics for equivalent household populations as well as pediatric kidney, heart, liver, lung transplant recipients and waitlisted patients.

DETAILED DESCRIPTION:
Influenza infections are a significant concern for the clinical management of transplant recipients, a highly vulnerable immunocompromised patient group. Early Influenza detection has major benefits for the successful treatment in that crucial early infection time window and allows for more timely mitigation measures to be employed. Xofluza® (Baloxavir Marboxil), FDA approved in 2018 for the treatment of acute Influenza, has been shown to have improved outcome characteristics versus Tamiflu® (Oseltamivir), as well as compliance (a single pill given once, versus 10 pills taken over 5 days for Oseltamivir). The timing of the influenza diagnoses and intervention greatly impacts the outcomes in both antiviral medications though. Smart wearable devices have demonstrated clear utility to detect early infection using physiological signatures such as sub-symptomatic increases in heart rate (HR) and body temperature. Detection of Influenza and severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) have been shown to be robustly detectable several days prior to clinical symptoms onset in large well-powered smartwatch studies.

This is a sub-study of the existing Institutional Review Board (IRB) # 20-017872 protocol: "Early Detection of SARS-CoV-2 & other Infections using Wearable Devices in Pediatric Transplant Patients and Household Members". This is a prospective, interventional, single-center study at The Children's Hospital of Philadelphia comprising kidney, heart, liver and lung transplant recipients, waitlisted patients, and their household members. Subjects will wear smart wearable devices to monitor biometrics including HR, HR variation (HRV) and proxies of body temperature. A smart wearable device alert generated from a validated early infection detection algorithm and alerting platform, precipitates subjects to use an at-home collection kit for SARS-CoV-2, Influenza A/B and respiratory syncytial virus (RSV) A/B which is then sent to a central clinical lab for polymerase chain reaction (PCR)-based diagnoses. If the transplant recipient is positive for Influenza A/B the local clinical care team will be informed to determine if Baloxavir and/or any other medication is warranted. Genentech will make the Baloxavir medication available via the CHOP transplant pharmacist through the recipients' regular pharmacy. If the non-transplanted household members are positive for Influenza or exposed to Influenza positive infected subject(s) their treatment will be determined by their own primary-care. All CHOP transplant recipients will have their medical records reviewed for relevant covariates and confounders after Baloxavir treatment. Study subjects will complete short daily REDCap symptom forms for the pre-, peri- and post-infection periods.

ELIGIBILITY:
Inclusion Criteria

Population 1: Potential Baloxavir treatment group (CHOP transplant subjects 5 years & up)

* Willing CHOP male or female kidney, heart, liver or lung single or multiple transplant recipients aged 5 years or older as per FDA guidelines.
* Willing to regularly wear a smartwatch and take an at-home positive respiratory virus (RV) panel which will include a diagnoses of Influenza A or B.
* Have an antigen positive diagnoses of Influenza A or B (a PCR-based positive clinical diagnoses of Influenza A or B may be requested in "alarm positive plus antigen positive but asymptomatic" cases).
* Can be included if their treating physician prescribe prophylactic treatment of Baloxavir if the subject has been exposed to Influenza.
* If Baloxavir is prescribed the study subject should be treated within 48 hours of symptom onset (regardless of the alarming time).

Population 2: Potential Baloxavir treatment group (CHOP waitlisted subjects 5 years & up)

• Willing waitlisted CHOP kidney, heart, liver or lung single or multiple transplant recipients aged 5 years or older, which are anticipated to have a transplant in the next 12 months.

Population 3: Potential Baloxavir treatment group (non-transplanted household members)

* Non-transplanted household member of a CHOP transplant recipient or waitlisted patient
* Be at least 5 years of age.
* Willing to regularly wear a smartwatch and take an at-home positive respiratory virus (RV) panel for diagnoses of Influenza A or B.
* Have a Antigen-based positive diagnoses of Influenza A or B

Population 4: Non-Baloxavir treatment subjects

* CHOP transplant recipients and all other non-transplanted household members who are 2-4 years of age.
* Subjects 5 years and up who are Influenza positive but whom do not receive Baloxavir treatment

Exclusion Criteria

Population 1:

* Any allergy to Baloxavir (although they can remain in the study as an influenza case or control without Baloxavir treatment, or if they have been treated with a different medication for influenza) or a recommendation from the study physicians'/transplant pharmacist(s) not to take Baloxavir.
* Subjects weighing < 20 kg
* If the subject is unable or unwilling to consent.
* If the subject is younger than 5 years of age.
* If the subject requires mechanical ventilation at time of enrollment.
* If the subject is pregnant or breast feeding at the time of early infection alerting.
* If the subject is taking a prohibited medication. These include Influenza antiviral drugs with the exception of oseltamivir and baloxavir (such as peramivir, laninamivir, zanamivir, rimantadine, umifenovir or amantadine).
* Unwilling or unable to comply with the study requirements.

Population 2: All exclusion criteria listed for Population 1

Population 3:

* Subjects weighing < 20 kg
* A household transplant recipient is not participating in the study
* Any allergy to Baloxavir (although they will remain in the study as an influenza case/control without treatment)
* A recommendation from the study physicians'/transplant pharmacist not to take Baloxavir
* If the subject is unable or unwilling to consent.
* If the subject is younger than 5 years of age.
* If the subject is pregnant at screening.
* If the subject is taking a prohibited medication. These include Influenza antiviral drugs with the exception of oseltamivir and baloxavir (such as peramivir, laninamivir, zanamivir, rimantadine, umifenovir or amantadine).
* Unwilling or unable to comply with the study requirements.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Time-to-Clinical-Response | 30 days post-Baloxavir treatment
  For subjects infected with Influenza investigators will assess Time-to-Clinical-Response in a time frame up to 30 days post Baloxavir treatment in this study vs comparable data available from national control groups. Time to Clinical Response is based on: (a) temperature ranges as measured by (standard of care and/or smartwatch biometric data), oxygen saturation, respiratory status, HR, and hospitalization status; (b) return to healthy baseline data including from biometric data derived from the subjects' smartwatch; (c) time to symptom resolution in a time frame up to 30 days post Baloxavir treatment as assessed from a return to healthy baseline on the daily questionnaires).
Incidence of complicated hospital stay(s) | 30 days post-Baloxavir treatment
  Incidence of complicated hospital stay(s) for a time frame up to 30 days post Baloxavir treatment in this study versus comparable data available from the previously described national control groups. A complicated hospital stay is defined as a hospital admission that was either prolonged (greater than 7 days), requiring ICU level of care or death at day 30 as a result of influenza infection.

SECONDARY OUTCOMES:
Incidence of Respiratory Tract Infection Progression Following Treatment | 30 days post-Baloxavir treatment
  Progression to lower respiratory tract infections in a time frame up to 30 days post Baloxavir treatment in this study versus comparable data available from national control groups.
Length of hospital Stay Following Treatment | 30 days post-Baloxavir treatment
  Length of hospital stay in a time frame up to 30 days post Baloxavir treatment in our study versus comparable data available from national control groups.
Oxygen requirement Following Treatment | 30 days post-Baloxavir treatment
  Oxygen requirement in a time frame up to 30 days post Baloxavir treatment in this study versus comparable data available from national control groups.
Rate of Respiratory Failure Following Treatment | 30 days post-Baloxavir treatment
  Rate of respiratory failure in a time frame up to 30 days post Baloxavir treatment in this study versus comparable data available from national control groups.
30-day Mortality Rate Following Treatment | 30 days post-Baloxavir treatment
  30-day mortality for post Baloxavir treatment in this study versus comparable data available from national control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew O Connor, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Summary-level statistics and outcomes of primary and secondary study endpoints will be made available to any study publications.

REFERENCES:
- [Background] Baxter D. Evaluating the case for trivalent or quadrivalent influenza vaccines. Hum Vaccin Immunother. 2016 Oct 2;12(10):2712-2717. doi: 10.1080/21645515.2015.1091130. Epub 2016 Jul 19. PMID 27435025
- [Background] Vanderlinden E, Naesens L. Emerging antiviral strategies to interfere with influenza virus entry. Med Res Rev. 2014 Mar;34(2):301-39. doi: 10.1002/med.21289. Epub 2013 Jun 25. PMID 23801557
- [Background] Tsang TK, Lau LLH, Cauchemez S, Cowling BJ. Household Transmission of Influenza Virus. Trends Microbiol. 2016 Feb;24(2):123-133. doi: 10.1016/j.tim.2015.10.012. Epub 2015 Nov 21. PMID 26612500
- [Background] Paules C, Subbarao K. Influenza. Lancet. 2017 Aug 12;390(10095):697-708. doi: 10.1016/S0140-6736(17)30129-0. Epub 2017 Mar 13. PMID 28302313
- [Background] Lee N, Ison MG. Diagnosis, management and outcomes of adults hospitalized with influenza. Antivir Ther. 2012;17(1 Pt B):143-57. doi: 10.3851/IMP2059. Epub 2012 Feb 3. PMID 22311561
- [Background] Kumar D, Michaels MG, Morris MI, Green M, Avery RK, Liu C, Danziger-Isakov L, Stosor V, Estabrook M, Gantt S, Marr KA, Martin S, Silveira FP, Razonable RR, Allen UD, Levi ME, Lyon GM, Bell LE, Huprikar S, Patel G, Gregg KS, Pursell K, Helmersen D, Julian KG, Shiley K, Bono B, Dharnidharka VR, Alavi G, Kalpoe JS, Shoham S, Reid GE, Humar A; American Society of Transplantation H1N1 Collaborative Study Group. Outcomes from pandemic influenza A H1N1 infection in recipients of solid-organ transplants: a multicentre cohort study. Lancet Infect Dis. 2010 Aug;10(8):521-6. doi: 10.1016/S1473-3099(10)70133-X. Epub 2010 Jul 9. PMID 20620116
- [Background] Kumar D, Ferreira VH, Blumberg E, Silveira F, Cordero E, Perez-Romero P, Aydillo T, Danziger-Isakov L, Limaye AP, Carratala J, Munoz P, Montejo M, Lopez-Medrano F, Farinas MC, Gavalda J, Moreno A, Levi M, Fortun J, Torre-Cisneros J, Englund JA, Natori Y, Husain S, Reid G, Sharma TS, Humar A. A 5-Year Prospective Multicenter Evaluation of Influenza Infection in Transplant Recipients. Clin Infect Dis. 2018 Oct 15;67(9):1322-1329. doi: 10.1093/cid/ciy294. PMID 29635437
- [Background] Noshi T, Kitano M, Taniguchi K, Yamamoto A, Omoto S, Baba K, Hashimoto T, Ishida K, Kushima Y, Hattori K, Kawai M, Yoshida R, Kobayashi M, Yoshinaga T, Sato A, Okamatsu M, Sakoda Y, Kida H, Shishido T, Naito A. In vitro characterization of baloxavir acid, a first-in-class cap-dependent endonuclease inhibitor of the influenza virus polymerase PA subunit. Antiviral Res. 2018 Dec;160:109-117. doi: 10.1016/j.antiviral.2018.10.008. Epub 2018 Oct 11. PMID 30316915
- [Background] O'Hanlon R, Shaw ML. Baloxavir marboxil: the new influenza drug on the market. Curr Opin Virol. 2019 Apr;35:14-18. doi: 10.1016/j.coviro.2019.01.006. Epub 2019 Mar 8. PMID 30852344
- [Background] Watanabe A, Ishida T, Hirotsu N, Kawaguchi K, Ishibashi T, Shishido T, Sato C, Portsmouth S, Tsuchiya K, Uehara T. Baloxavir marboxil in Japanese patients with seasonal influenza: Dose response and virus type/subtype outcomes from a randomized phase 2 study. Antiviral Res. 2019 Mar;163:75-81. doi: 10.1016/j.antiviral.2019.01.012. Epub 2019 Jan 23. PMID 30684563
- [Background] Hayden FG, Sugaya N, Hirotsu N, Lee N, de Jong MD, Hurt AC, Ishida T, Sekino H, Yamada K, Portsmouth S, Kawaguchi K, Shishido T, Arai M, Tsuchiya K, Uehara T, Watanabe A; Baloxavir Marboxil Investigators Group. Baloxavir Marboxil for Uncomplicated Influenza in Adults and Adolescents. N Engl J Med. 2018 Sep 6;379(10):913-923. doi: 10.1056/NEJMoa1716197. PMID 30184455
- [Background] Ison MG, Portsmouth S, Yoshida Y, Shishido T, Mitchener M, Tsuchiya K, Uehara T, Hayden FG. Early treatment with baloxavir marboxil in high-risk adolescent and adult outpatients with uncomplicated influenza (CAPSTONE-2): a randomised, placebo-controlled, phase 3 trial. Lancet Infect Dis. 2020 Oct;20(10):1204-1214. doi: 10.1016/S1473-3099(20)30004-9. Epub 2020 Jun 8. PMID 32526195
- [Background] Baker J, Block SL, Matharu B, Burleigh Macutkiewicz L, Wildum S, Dimonaco S, Collinson N, Clinch B, Piedra PA. Baloxavir Marboxil Single-dose Treatment in Influenza-infected Children: A Randomized, Double-blind, Active Controlled Phase 3 Safety and Efficacy Trial (miniSTONE-2). Pediatr Infect Dis J. 2020 Aug;39(8):700-705. doi: 10.1097/INF.0000000000002747. PMID 32516282
- [Background] Ikematsu H, Hayden FG, Kawaguchi K, Kinoshita M, de Jong MD, Lee N, Takashima S, Noshi T, Tsuchiya K, Uehara T. Baloxavir Marboxil for Prophylaxis against Influenza in Household Contacts. N Engl J Med. 2020 Jul 23;383(4):309-320. doi: 10.1056/NEJMoa1915341. Epub 2020 Jul 8. PMID 32640124
- [Background] Umemura T, Mutoh Y, Kawamura T, Saito M, Mizuno T, Ota A, Kozaki K, Yamada T, Ikeda Y, Ichihara T. Efficacy of baloxavir marboxil on household transmission of influenza infection. J Pharm Health Care Sci. 2020 Oct 1;6:21. doi: 10.1186/s40780-020-00178-4. eCollection 2020. PMID 33014405
- [Background] Shirley M. Baloxavir Marboxil: A Review in Acute Uncomplicated Influenza. Drugs. 2020 Jul;80(11):1109-1118. doi: 10.1007/s40265-020-01350-8. PMID 32601915
- [Background] Neuberger E, Wallick C, Chawla D, Castro RC. Baloxavir vs oseltamivir: reduced utilization and costs in influenza. Am J Manag Care. 2022 Mar 1;28(3):e88-e95. doi: 10.37765/ajmc.2022.88786. PMID 35404552
- [Background] Alavi A, Bogu GK, Wang M, Rangan ES, Brooks AW, Wang Q, Higgs E, Celli A, Mishra T, Metwally AA, Cha K, Knowles P, Alavi AA, Bhasin R, Panchamukhi S, Celis D, Aditya T, Honkala A, Rolnik B, Hunting E, Dagan-Rosenfeld O, Chauhan A, Li JW, Bejikian C, Krishnan V, McGuire L, Li X, Bahmani A, Snyder MP. Real-time alerting system for COVID-19 and other stress events using wearable data. Nat Med. 2022 Jan;28(1):175-184. doi: 10.1038/s41591-021-01593-2. Epub 2021 Nov 29. PMID 34845389
- [Background] Keating BJ, Mukhtar EH, Elftmann ED, Eweje FR, Gao H, Ibrahim LI, Kathawate RG, Lee AC, Li EH, Moore KA, Nair N, Chaluvadi V, Reason J, Zanoni F, Honkala AT, Al-Ali AK, Abdullah Alrubaish F, Ahmad Al-Mozaini M, Al-Muhanna FA, Al-Romaih K, Goldfarb SB, Kellogg R, Kiryluk K, Kizilbash SJ, Kohut TJ, Kumar J, O'Connor MJ, Rand EB, Redfield RR, Rolnik B, Rossano J, Sanchez PG, Alavi A, Bahmani A, Bogu GK, Brooks AW, Metwally AA, Mishra T, Marks SD, Montgomery RA, Fishman JA, Amaral S, Jacobson PA, Wang M, Snyder MP. Early detection of SARS-CoV-2 and other infections in solid organ transplant recipients and household members using wearable devices. Transpl Int. 2021 Jun;34(6):1019-1031. doi: 10.1111/tri.13860. Epub 2021 May 5. PMID 33735480
- [Background] Mishra T, Wang M, Metwally AA, Bogu GK, Brooks AW, Bahmani A, Alavi A, Celli A, Higgs E, Dagan-Rosenfeld O, Fay B, Kirkpatrick S, Kellogg R, Gibson M, Wang T, Hunting EM, Mamic P, Ganz AB, Rolnik B, Li X, Snyder MP. Pre-symptomatic detection of COVID-19 from smartwatch data. Nat Biomed Eng. 2020 Dec;4(12):1208-1220. doi: 10.1038/s41551-020-00640-6. Epub 2020 Nov 18. PMID 33208926
- [Background] Grzesiak E, Bent B, McClain MT, Woods CW, Tsalik EL, Nicholson BP, Veldman T, Burke TW, Gardener Z, Bergstrom E, Turner RB, Chiu C, Doraiswamy PM, Hero A, Henao R, Ginsburg GS, Dunn J. Assessment of the Feasibility of Using Noninvasive Wearable Biometric Monitoring Sensors to Detect Influenza and the Common Cold Before Symptom Onset. JAMA Netw Open. 2021 Sep 1;4(9):e2128534. doi: 10.1001/jamanetworkopen.2021.28534. PMID 34586364
- [Background] Vilchez RA, McCurry K, Dauber J, Lacono A, Griffith B, Fung J, Kusne S. Influenza virus infection in adult solid organ transplant recipients. Am J Transplant. 2002 Mar;2(3):287-91. doi: 10.1034/j.1600-6143.2002.20315.x. PMID 12096793
- [Background] Marois C, Nedelec T, Pelle J, Rozes A, Durrleman S, Dufouil C, Demoule A. Comparison of Clinical Profiles and Mortality Outcomes Between Influenza and COVID-19 Patients Invasively Ventilated in the ICU: A Retrospective Study From All Paris Public Hospitals From 2016 to 2021. Crit Care Explor. 2022 Jul 25;4(7):e0737. doi: 10.1097/CCE.0000000000000737. eCollection 2022 Jul. PMID 35923591
- [Background] Helantera I, Gissler M, Rimhanen-Finne R, Ikonen N, Kanerva M, Lempinen M, Finne P. Epidemiology of laboratory-confirmed influenza among kidney transplant recipients compared to the general population-A nationwide cohort study. Am J Transplant. 2021 May;21(5):1848-1856. doi: 10.1111/ajt.16421. Epub 2021 Feb 19. PMID 33252189
- [Background] Mombelli M, Kampouri E, Manuel O. Influenza in solid organ transplant recipients: epidemiology, management, and outcomes. Expert Rev Anti Infect Ther. 2020 Feb;18(2):103-112. doi: 10.1080/14787210.2020.1713098. Epub 2020 Jan 18. PMID 31910344
- [Background] Kuchipudi SV, Behring D, Nissly R, Chothe SK, Gontu A, Ravichandran A, Butler T. Mitigating the Impact of Emerging Animal Infectious Disease Threats: First Emerging Animal Infectious Diseases Conference (EAIDC) Report. Viruses. 2022 Apr 30;14(5):947. doi: 10.3390/v14050947. PMID 35632689